CLINICAL TRIAL: NCT00236223
Title: The Effect of Gabapentin, Low Dose Ketamine, Paracetamol, NSAID and Dexamethasone on Pain and Opioid Requirements in Patients Scheduled for Primary Total Hip Replacement
Brief Title: The Effect of Gabapentin, Ketamine and Dexamethasone on Pain and Opioid Requirements After Hip Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Structural changes that stopped the type of operations used in the study
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Ole Mathiesen, Dept of anaesthesiology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM2-05
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2008-05-15 (Estimated); Status verified 2008-05

CONDITIONS: Pain, Postoperative
Keywords: Primary hip replacement; Gabapentin; Dexamethasone; Ketamine; Multimodal postoperative analgesia.
MeSH Terms: conditions — Pain, Postoperative | interventions — Gabapentin; Dexamethasone; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Gabapentin + dexamethasone + ketamine
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin + dexamethasone + ketamine — Comparing analgesic effect of gabapentin 1200 mg + dexamethasone 8 mg + ketamine 0.15 mg/kg
  Other Names: Anti-hyperalgesics; Postoperative pain
  Arms: 1
Drug: Placebo — Matching placebo
  Arms: 2

SUMMARY:
Patients scheduled for primary hip replacement needs postoperative pain treatment, i.e. morphine. Morphine has side-effects: nausea, vomiting, sedation and dizziness. These side-effects are unpleasant for the patients and sometimes keeps them at bed longer time than needed. We investigate in new combinations of analgesics for postoperative pain, hoping to minimize the need for morphine.

DETAILED DESCRIPTION:
The effect on postoperative pain of the combination of preoperative gabapentin 1200 mg + dexamethasone 8 mg + ketamine 0.15mg/kg versus placebo is investigated on patients having a hip alloplastic operation.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for primary total hip replacement,
* Between 55 and 85 years of age,
* ASA 1-3 and BMI between 18 and 35.

Exclusion Criteria:

Patients who are:

* Unable to cooperate
* Does not speak Danish
* Has allergy for drugs used in the trial
* Drug or alcohol abuse
* Epilepsy
* Medically treated diabetes
* Known kidney disease
* Daily use of analgetics
* Apart from NSAID
* Paracetamol or COX2 inhibitors
* Are treated with a antidepressive.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-10; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The total amount of morphine needed postoperatively from 0-4h; and 0-24h, administered by a patient controlled pain treatment.(PCA) | 0-24h

SECONDARY OUTCOMES:
Pain score (VAS)= at rest and at mobilisation. | 0-24h
Postoperative Nausea and vomiting. | 0-24h
Dizziness | 0-24h
Sedation | 0-24h
Nightmare and hallucinations. | 0-24h
All measurements are taken at 2,4 and 24 h postoperatively. | 0-24h

CONTACTS AND LOCATIONS:
Overall Officials: Ole Mathiesen, MD, Principal Investigator — Department of Anaesthesiology, Copenhagen University Hospital in Glostrup, 2600 Glostrup, Denmark
Locations (2):
- Denmark (2):
  - Operations og Anæstesiologisk afd. Y, KAS Glostrup, Glostrup Municipality
  - Anæstesiafdelingen, Herning Centralsygehus, Herning